CLINICAL TRIAL: NCT02289872
Title: Comparison of the TruView PCD Video Laryngoscope and Macintosh Laryngoscope for Pediatric Tracheal Intubation by Novice Paramedics: A Randomized Crossover Simulation Trial.
Brief Title: Pediatric Intubation
Acronym: ETICPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TruView/01
Record Dates: First submitted 2014-11-07; First posted 2014-11-13 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Intubation; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Scenario A (Experimental): The control scenario, where neither chest compression nor cervical stabilization was applied during intubation.
  Interventions: Device: Macintosh Laryngoscope; Device: TruView PCD Video laryngoscope
- Scenario B (Experimental): The chest compression scenario, where continuous chest compression was applied using chest compression system LUCAS-2 (Physio-Control, Redmond, WA, USA). Chest compression was provided at a rate of 100 min-1 to a depth of 5-6 cm during all intubation procedures.
  Interventions: Device: Macintosh Laryngoscope; Device: TruView PCD Video laryngoscope
- Scenario C (Experimental): The chest compression with cervical stabilization scenario, where both chest compression using Lucas-2 and cervical stabilization were applied. A correctly fitting standard cervical immobilization collar (StifNeck Select, Laerdal, Stavanger, Norway) was applied to the manikin's neck to prevent movement of the cervical spine.
  Interventions: Device: Macintosh Laryngoscope; Device: TruView PCD Video laryngoscope

INTERVENTIONS:
Device: Macintosh Laryngoscope — Direct-Laryngoscopy
Device: TruView PCD Video laryngoscope — Video-Laryngoscopy

SUMMARY:
The aim of the study was to compare time and success rates of TruView PCD video laryngoscope and Macintosh laryngoscope for the pediatric emergency intubation with three airway scenarios in a standardized manikin model.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* inexperienced in pediatric intubation paramedics

Exclusion Criteria:

* not meet the above criteria
* participants who had performed intubation in pediatric humans prior the trial or had previously TruView experience

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to intubation | 1 day
  the time to intubation, defined as the time from insertion of the laryngoscope blade between the teeth to the first manual ventilation of the mannequin's lungs

SECONDARY OUTCOMES:
Success of intubation | 1 day
  success of the intubation attempt (i.e. tracheal or oesophageal placement of the tube) with was recorded when the success of the ventilation attempt was seen by the manikin's ventilation indicators.
Cormack-Lehan scale | 1 day
  self reported Cormack-Lehan scale during intubation
Dental compression | 1day
  dental compression, with was assessed using a visual scale grading the pressure applied on the upper teeth (n=none, mild=1, moderate=2, severe=3).
Ease of intubation (VAS) | 1 day
  To access subjective opinion about the difficulty of the each intubation method, participants were asked to rate it on a visual analogue scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult).

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovie, Poland

REFERENCES:
- [Derived] Szarpak L, Czyzewski L, Kurowski A, Truszewski Z. Comparison of the TruView PCD video laryngoscope and macintosh laryngoscope for pediatric tracheal intubation by novice paramedics: a randomized crossover simulation trial. Eur J Pediatr. 2015 Oct;174(10):1325-32. doi: 10.1007/s00431-015-2538-0. Epub 2015 Apr 18. PMID 25894914